CLINICAL TRIAL: NCT06788405
Title: Development of Hand Hygiene Training Virtual Reality Simulation and Evaluation of Its Effectiveness: an Example of In-Service Training in Nursing
Brief Title: Development of Hand Hygiene Training Virtual Reality Simulation and Evaluation of Its Effectiveness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Askin Selvi, Nurse Educator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: İUC_ASELVİ_001; Hülya Kaya (Other: Bezm-i Alem Foundation University)
Record Dates: First submitted 2024-04-12; First posted 2025-01-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hospital Infection
Keywords: hand hygiene; virtual reality; nursing education
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Other: hand hygiene theoretical training with a hand hygiene virtual reality simulation application
- control group (Other)
  Interventions: Other: hand hygiene theoretical training

INTERVENTIONS:
Other: hand hygiene theoretical training with a hand hygiene virtual reality simulation application — After giving 360 hours of hand hygiene theoretical training to the participants in the experimental group, a hand hygiene virtual reality simulation application will be performed.
  Arms: experimental group
Other: hand hygiene theoretical training — Participants in the control group will receive only 360 hours of hand hygiene theoretical training. Participants in this group will not be given hand hygiene virtual reality simulation application.
  Arms: control group

SUMMARY:
Healthcare-associated infections (HAI), which have become a major problem in all countries, prolong hospital stay and increase treatment and care costs. In health care institutions, HAIs that occur directly or indirectly related to health services are among the most common causes of mortality and morbidity. A high level of hand hygiene compliance, which is the most basic step of infection control and precautions, is the first and most important step to prevent HAIs. However, it has been determined in the literature that the compliance rates of healthcare professionals with hand hygiene are low and that nurses' attitudes and behaviors regarding hand hygiene are not at the desired level. Well-structured training programs need to be developed to maintain and increase nurses' hand hygiene compliance rates. Different training methods and tools are needed to increase hand hygiene compliance, awareness and awareness. It is recommended that innovative training approaches such as virtual simulation be developed and evaluated to further internalize and encourage nurses' most effective hand hygiene practice behaviors. In recent years, the use of simulation methods in the training of healthcare professionals has been increasing as they facilitate the transfer of theoretical knowledge into clinical practice. One of these simulation methods is virtual reality (VR). The use of gamification in the virtual environment supports different learning styles, enabling learners to participate more intensively in education and increase their internal motivation. In this context, with VR support, entertainment and learning processes can be used to support each other. Considering the features of VR usage such as integrating knowledge and skills, creating a learning environment for the learner by doing, giving the opportunity to repeat until the correct application is made, reducing incorrect interventions in clinical practice and increasing patient safety, it is recommended that virtual simulation systems be used in nursing education. VR provides different opportunities to learners by enriching and diversifying learning environments. In these virtual environments, learners can have new experiences and these experiences remain permanent for the learners. As stated in the WHO Hand Hygiene Theme, it is important to develop innovative training programs, learning materials and measurement and evaluation tools regarding hand hygiene within the scope of infection control and prevention studies. VR simulation can be used to attract nurses' attention and awareness by increasing intrinsic motivation to perform hand hygiene, and can be used to support nurses in developing positive attitudes towards hand hygiene. Hand hygiene simulation scenarios created with virtual reality can contribute to greater awareness about the problems caused by microorganism transmission by increasing hand hygiene awareness. Thus, increasing attitudes and awareness regarding hand hygiene can have a positive effect on reducing the HAI rate by supporting the transformation of hand hygiene awareness into behavior. In the study, it was planned to develop, implement and evaluate a virtual reality hand hygiene simulation. It is thought that this virtual reality simulation will pave the way for the development of psychomotor skills for hand hygiene, increase the level of knowledge, and increase hand hygiene compliance by providing internal motivation to perform hand hygiene. In our country, no studies have been found on the development of virtual reality simulation in hand hygiene practice. The aim of this study is to develop and implement virtual reality hand hygiene simulation in teaching hand hygiene behaviors in nurses and to evaluate its effect on hand hygiene compliance.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who have not received additional hand hygiene training after general orientation training at the beginning of work • Nurses working actively in areas other than the operating room (inpatient services, intervention units, etc.).

Exclusion Criteria:

* Nurses in the intervention group who have a disease/condition that may pose a problem regarding the use of VR glasses (having epilepsy, having a history of seizures, having an eye or neurological disease that would prevent the use of VR glasses, having motion sickness).

  * Nurses working in the operating room
  * Nurses who receive additional hand hygiene training after general orientation training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Introductory Form | up to one month
  It is an introductory form prepared by the researcher as a result of a literature review, which includes questions about the socio-demographic characteristics of the participants, their current situation in the working environment regarding hand hygiene, and their opinions about hand hygiene.
Knowledge Test | up to 12 weeks
  It is a form prepared by the researcher after a literature review to evaluate the level of knowledge about hand hygiene to be applied before and after hand hygiene training and will be used after validity and reliability analysis.
Scale for Evaluation of Hand Washing Behavior in Terms of Planned Behavior Model | up to 12 weeks
  The scale was developed to collect information about the knowledge, attitudes and behaviors of healthcare personnel regarding hand washing and to identify deficiencies. The scale consists of 8 sub-dimensions and a total of 46 items related to knowledge, attitudes and behaviors towards hand washing. The lowest score that can be obtained from the scale is 46, the highest score is 176. A high score indicates a positive and strong motivation to wash hands.
Hand Hygiene Observation Form | up to 12 weeks
  This form is prepared with reference to the World Health Organization and is marked by observing hand hygiene behaviors in clinics. In the Hand Hygiene Observation Form, the observed indications are classified as the appropriate time for hand hygiene (denominator) used to measure the actual hand hygiene action (action serving as the numerator). These two variables determine the compliance to be calculated. Compliance results can be calculated overall, but can also be divided into occupational categories and indications. Compliance with hand hygiene is the ratio of the number of actions to the number of appropriate times and is expressed by the following formula:
  Compliance (%) = Number of WASHES and/or SCRUBS × 100 / Number of Indications
  Compliance by Indication (%) = Number of WASHES and/or SCRUBS × 100 / Number of Indications
Simulation Design Scale | up to 12 weeks
  The scale is evaluated in 2 parts. In the first part; It is evaluated whether the best simulation design elements can be applied in the simulation application. In the second part; It evaluates how important the simulation design elements are for the participants. The first section is evaluated as "strongly disagree with the statement", "disagree with the statement", "undecided", "agree with the statement", "strongly agree with the statement" and "not appropriate". The second section is evaluated as "not important", "partially important", "undecided", "important", "very important". Scale scores are obtained by dividing the sum of the total and sub-dimension scores by the number of items.
Training Evaluation Form | up to 12 weeks
  It is a form prepared for participants to evaluate the purpose of the training program, training activities, satisfaction level with the program, training environment and educator. It is not a scale, but a form prepared by the researcher.
Student Satisfaction and Self-Confidence Scale in Learning | up to 12 weeks
  It is a scale that determines the satisfaction level of the participants towards the simulation application. Scale scores are obtained by dividing the total of the sub-dimensions by the number of items. As the total score from the scale increases, student satisfaction and self-confidence in learning also increase.

CONTACTS AND LOCATIONS:
Overall Officials: AŞKIN SELVİ, PhD student, Principal Investigator — İstanbul University-Cerrahpasa, Turkey
Locations (1):
- Aşkin Selvi, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol Statistical Analysis Plan Informed Consent Form Clinical Study Report Analytic Code

REFERENCES:
- [Background] Clack, L., Hirt, C., Kunz, A., Sax, H. 2021. "Experiential training of hand hygiene using virtual reality. recent advances in technologies for ınclusive well-being", 196: 31-42. Doi: 10.1007/978-3-030-59608-8_3.
- [Background] Eichel VM, Brandt C, Brandt J, Jabs JM, Mutters NT. Is virtual reality suitable for hand hygiene training in health care workers? Evaluating an application for acceptability and effectiveness. Antimicrob Resist Infect Control. 2022 Jun 25;11(1):91. doi: 10.1186/s13756-022-01127-6. PMID 35752839